CLINICAL TRIAL: NCT03336021
Title: Impact Evaluation of Agribusiness Support and Nutrition Services Projects in Upper Egypt
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Intervention not implemented as planned
Sponsor: International Food Policy Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 602114.002.001
Record Dates: First submitted 2017-10-26; First posted 2017-11-08 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2017-11

CONDITIONS: Poverty, Low Income, Food Insecurity, Undernutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Enumerators will be blinded (to the extent possible) to the treatment assignment of farmers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): FAS program
  Interventions: Other: FAS program
- Comparison (No Intervention): Comparison group

INTERVENTIONS:
Other: FAS program — Intervention households are farmers who will receive a forward contract through the FAS program; in addition, they may receive other support such as extension, seeds, etc.
  Arms: Intervention

SUMMARY:
This project seeks to evaluate the impact of two USAID-funded projects that are implemented in rural Upper Egypt. The first project is the Feed the Future Egypt, Food-Security and Agribusiness Support (FAS) project; the second project is the Improving Maternal, Child Health, and Nutrition Services (IMCHN) project.

The specific study objectives are (1) to estimate the impact of FAS interventions on project outcome indicators-especially on household income (measured by total household expenditure), household food security, and maternal and child nutrition-among farm households; (2) to estimate the effects of IMCHN interventions on maternal and child health and nutrition knowledge among community health workers (CHWs) and among farm households; and (3) to analytically explore potential synergistic effects of FAS and IMCHN interventions on maternal and child nutrition among farm households being exposed to both projects.

ELIGIBILITY:
Inclusion Criteria (will follow those of the USAID-funded FAS program). In Oct 2017, known to be:

* Farmers with 10 feddans or less per household
* Farmers who have experience or interest in horticulture production.

Exclusion Criteria:

* Farmers with more than 10 feddans per household
* Farmers with no interest in horticulture production

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Household income | After 5 to 6 months of exposure (april 2018)
  household income measured through household total (and food) expenditure
Household food security | After 5 to 6 months of exposure (april 2018)
  Household Food Insecurity Access Scale (HFIAS)

SECONDARY OUTCOMES:
Household income | After 17 to 18 months of exposure (april 2019)
  household income measured through household total (and food) expenditure
Household food security | After 17 to 18 months of exposure (april 2019)
  Household Food Insecurity Access Scale (HFIAS)
Farm production and output: yields | After 5 to 6 months of exposure (april 2018) and after 17 to 18 months of exposure (april 2019)
  Harvested yields
Farm production and output: prices | After 5 to 6 months of exposure (april 2018) and after 17 to 18 months of exposure (april 2019)
  Selling prices
Farm production and output: home consumption | After 5 to 6 months of exposure (april 2018) and after 17 to 18 months of exposure (april 2019)
  Home consumption
Women's Empowerment in Agriculture | After 5 to 6 months of exposure (april 2018) and after 17 to 18 months of exposure (april 2019)
  Women's level of empowerment in agriculture-related decision making
Household dietary diversity | After 5 to 6 months of exposure (april 2018) and after 17 to 18 months of exposure (april 2019)
  Household Dietary Diversity Score (HDDS)
Women's dietary diversity | After 5 to 6 months of exposure (april 2018) and after 17 to 18 months of exposure (april 2019)
  Minimum Dietary Diversity - Women (MDD-W) score
Infant and Young Child Feeding practices | After 5 to 6 months of exposure (april 2018) and after 17 to 18 months of exposure (april 2019)
  IYCF practices as measured using the WHO IYCF guidelines
Child anthropometry: weight | After 5 to 6 months of exposure (april 2018) and after 17 to 18 months of exposure (april 2019)
  weight of children 0-23.9 months (baseline), 24-59.9 months (baseline)
Child anthropometry: height | After 5 to 6 months of exposure (april 2018) and after 17 to 18 months of exposure (april 2019)
  height and weight of children 0-23.9 months (baseline), 24-59.9 months (baseline)
Adult anthropometry: mother | After 5 to 6 months of exposure (april 2018) and after 17 to 18 months of exposure (april 2019)
  weight of mother / female caretaker
Adult anthropometry: father | After 5 to 6 months of exposure (april 2018) and after 17 to 18 months of exposure (april 2019)
  weight of father / household head

OTHER OUTCOMES:
Nutrition and health knowledge of community health workers | After 5 to 6 months of exposure (april 2018) and after 17 to 18 months of exposure (april 2019)
  Community health workers' knowledge of nutrition and health related issues

CONTACTS AND LOCATIONS:
Overall Officials: Clemens Breisinger, PhD, Study Director — IFPRI; Jose Luis Figueroa, PhD, Principal Investigator — IFPRI

IPD SHARING:
Plan to Share IPD: Undecided